CLINICAL TRIAL: NCT02190474
Title: Mindfulness Interventions and Chronic Symptoms
Brief Title: Mindfulness Interventions and Chronic Widespread Pain in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1201009502; K23AT006703 (NIH)
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Fibromyalgia; Chronic Widespread Pain
Keywords: fibromyalgia; juvenile fibromyalgia; juvenile primary fibromyalgia syndrome (JPFS); adolescent pain; mindfulness; MBSR
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mindfulness Group (Experimental): These adolescents will be invited to participate in a group mindfulness meditation program based on a protocol refined by the investigative team. The weekly group meetings will be taught by an MBSR teacher at the Yale School of Medicine, with experience teaching mindfulness interventions to adults, children, and adolescents.
  Interventions: Behavioral: Mindfulness Group

INTERVENTIONS:
Behavioral: Mindfulness Group — Participants will attend weekly 1-2-hour group sessions (of 6-8 persons) led by a trained expert based on the working MBSR protocol. The weekly sessions will be scheduled in a time mutually convenient for participants and their parent/guardian that will accompany them to each group session. The MBSR group sessions will take place at the Yale School of Medicine.

SUMMARY:
The primary objective of this study to determine the feasibility and acceptability of a mindfulness intervention for adolescents with juvenile fibromyalgia/ chronic widespread pain and other similar chronic symptoms.

DETAILED DESCRIPTION:
The primary objective is to test the feasibility, safety, tolerability and acceptability of a mindfulness meditation intervention for adolescents with juvenile fibromyalgia/chronic widespread pain.

The purpose of the program is to test how effective an 8-week meditation and stress reduction class is in helping adolescents with chronic symptoms (including but not limited to fibromyalgia or chronic widespread pain, irritable bowel syndrome, joint pain, chronic fatigue, and others).

Participants will attend group sessions led by an instructor experienced in MBSR in an academic setting. The mindfulness meditation group sessions will take place at the Yale School of Medicine.

Participants will attend 90-minute weekly group sessions and a 4-hour retreat with approximately 6-8 other study participants at Yale School of Medicine. Participants are asked to practice at home by listening to pre-recorded 15-20 minute guided meditations.

ELIGIBILITY:
Inclusion Criteria:

* 2010 American College of Rheumatology (ACR) criteria based on the Widespread Pain Index (WPI) and Symptom Severity (SS) checklist.
* Functional Disability Score ≥13 indicating at least moderate disability
* Average pain intensity in the past week ≥ 4 on a 0-10 cm Visual Analog Scale.
* Access to mobile telephone/smartphone with text messaging plan in order to receive survey questions.
* Chronic symptoms such as fatigue, pain, bowel dysfunction, perceived cognitive impairment, or other non-specific symptoms persisting for 3-months or more, severe enough to have led to more than one visit to a medical provider. These symptoms must have not been found to be due to a definable general medical disorder despite adequate evaluation.

Exclusion Criteria:

* Diagnosis of an autoimmune or rheumatologic disease
* Current regular mindfulness meditation activity
* Serious illness (including mental illness/psychopathology) within 90 days prior to screening
* Inability or unwillingness of a parent to give consent/permission or child to assent
* Current use of opioid analgesics
* Current prescription for antidepressant medications
* Screening positive on the Columbia Suicide Screen (CSS)
* Active participation (weekly or more often) in a fibromyalgia or chronic disease support group

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2014-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Feasibility and retention | 8 weeks
  Feasibility and retention will be assessed after each cohort completes the group sessions. Feasibility of the intervention will be assessed by the proportion of eligible patients approached for the study who consent to participate and the proportion of the weekly sessions that are attended.

SECONDARY OUTCOMES:
Program Adherence | 8 weeks
  Program adherence will be tracked by assessing the actual amount of home practice in minutes per week using weekly self-report diaries.
Program Use | 8 weeks
  Program use will be assessed by quantifying the amount of minutes that participants spent practicing MBSR. Participants will agree to receive and respond to a daily question of "How many minutes did you spend practicing MBSR yesterday" delivered by SMS/text message to their mobile telephone.
Program Practicality | 8 weeks
  Program practicality will be qualitatively assessed. Practicality (ability to attend intervention sessions and practice at home), interest in the intervention, perceived effectiveness, will be collected through brief (15-20 min) interviews following completion of the 8-week intervention.
Functional Disability Inventory (FDI) | 8 weeks
  The FDI assesses functional disability (physical and psychosocial functional impairment) in children and adolescents with chronic pain. Scores range from 0-60, with higher scores indicating greater functional disability, categorized as No/Minimal (0-12), Moderate (13-29), and Severe (30) Disability.
Juvenile Revised Fibromyalgia/Symptom Impact Questionnaire (FIQR/SIQR) | 8 weeks
  The FIQR-C (and analogue SIQR) is a pediatric version of the adult Revised Fibromyalgia Impact Questionnaire that has been the major physical function assessment in adult fibromyalgia trials. The FIQR has credible construct validity, reliable test-retest characteristics and good sensitivity in demonstrating therapeutic change. The FIQR-C is used to measure subjects' physical function, overall impact of the syndrome, and symptom severity. It is scored from 0 (best) to 100 (worst) and takes less than 2 minutes to complete.
Pediatric Quality of Life Inventory (PedsQL) 4.0 (Adolescent Form) | 8 weeks
  PedsQL 4.0 (Pediatric Quality of Life Inventory) is a modular instrument for measuring health-related quality of life in children and adolescents ages 2 to 18. The PedsQL 4.0 Generic Core Scales are multidimensional child self-report and parent proxy-report scales developed as the generic core measure to be integrated with the PedsQL Disease-Specific Modules. The PedsQL 4.0 Generic Core Scales consist of 23 items applicable for healthy school and community populations, as well as pediatric populations with acute and chronic health conditions.
Perceived Stress Scale (PSS) | 8 weeks
  The PSS is a 14-item scale that assesses perceived stress of life situations in adolescents and adults. Items are scored on a 5-point scale (0=never to 4=very often). Higher total scores indicate greater levels of perceived stress. The PSS has well-established validity in relation to physiological stress responses, anxiety, and depressive disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Ather Ali, ND, MPH, MHS, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Result] Ali A, Weiss TR, Dutton A, McKee D, Jones KD, Kashikar-Zuck S, Silverman WK, Shapiro ED. Mindfulness-Based Stress Reduction for Adolescents with Functional Somatic Syndromes: A Pilot Cohort Study. J Pediatr. 2017 Apr;183:184-190. doi: 10.1016/j.jpeds.2016.12.053. Epub 2017 Jan 12. PMID 28088398